CLINICAL TRIAL: NCT03498040
Title: Development and Progression of Carcinoid Heart Disease in a Cohort of Adult Patients With Neuroendocrine Tumors Carcinoid Heart Disease (CHD): An Observational French Multi-Centre Cohort Study CRUSOE - NETs (CaRdiac UltraSonic OutcomEs - NETs)
Brief Title: Development and Progression of Carcinoid Heart Disease in a Cohort of Adult Patients With Neuroendocrine Tumors
Acronym: CRUSOE-NETs
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0700
Record Dates: First submitted 2018-03-23; First posted 2018-04-13 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Carcinoid Heart Disease
MeSH Terms: conditions — Carcinoid Heart Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with or at risk of carcinoid heart disease: * Adult patients with well-differentiated metastatic ileum or bronchial neuroendocrine tumor
  * Adult patients with carcinoid syndrome or elevated urinary 5HIAA regardless of primary site
  Interventions: Other: Study of the occurrence of Carcinoid Heart Disease

INTERVENTIONS:
Other: Study of the occurrence of Carcinoid Heart Disease — Patient at high risk of Carcinoid Heart Disease (metastatic ileum or bronchial well-differentiated neuroendocrine tumors, patients with high level of urinary 5HIAA or with carcinoid syndrome) are followed with annual echocardiography to detect the occurrence of carcinoid heart disease.
  In case of documented Carcinoid Heart Disease, a six or three months' cardiac follow-up is necessary to evaluate the progression and the severity of the disease.
  Investigators collect the data of clinical parameters (flushes, diarrhea, …) biological parameters (urinary 5HIAA, NT-ProBNP …) and cardiac parameters that may influence the occurrence, severity and progression of Carcinoid Heart Disease.

SUMMARY:
Carcinoid Heart Disease (CHD) is a rare form of heart disease, occurring in over 50% of the patients with carcinoid syndrome. Pathophysiology, prognostic factors of development of Carcinoid Heart Disease and progression of disease remain unclear.

This observational multicenter cohort study is designed to study the occurrence of Carcinoid Heart Disease in patients with differentiated carcinoid tumors, to describe numerous factors influencing the occurrence, severity, progression and long-term survival of patients with Carcinoid Heart Disease. Basic informations and detailed diagnosis informations (oncological and cardiac parameters), are collected by professional doctors. Clinical outcomes (onset of Carcinoid Heart Disease, cardiac surgery, related death) will be followed up every year or every six/three months if clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients followed in a NeuroEndocrine Tumor center with a reference cardiologist
* Patient with:

  * Histologically documented metastatic well-differentiated ileum neuroendocrine tumor or
  * Histologically documented metastatic well-differentiated bronchial neuroendocrine tumor, or
  * Histologically documented well differentiated neuroendocrine tumor, regardless of the primitive site or unknown primitive site and presenting a carcinoid syndrome and / or an elevation of urinary 5HIAA > 2 fold the upper limit of normal range
* Information given to the patient and his documented non-opposition

Exclusion Criteria:

* Poorly differentiated neuroendocrine carcinoma
* Patient unable / unwilling to follow the cardiac monitoring recommended by good practice data
* Any medical, geographical, sociological, psychological or legal situation that does not allow the patient to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with metastatic well-differentiated ileum or bronchial neuroendocrine tumor, adult patients with carcinoid syndrome and/or urinary 5HIAA > 2 fold the upper limit of normal regardless the primary site of the tumor, and therefore likely to develop Carcinoid Heart Disease (CHD).
Sampling Method: Non-Probability Sample
Enrollment: 670 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2033-04-16 (Estimated); Study Completion 2033-04-16 (Estimated)

PRIMARY OUTCOMES:
Carcinoid Heart Disease | 10 years (at the end of study)
  Percentage of patients with carcinoid heart disease at diagnosis and during follow-up (carcinoid heart disease diagnosis will be assessed by an annual echocardiography).

SECONDARY OUTCOMES:
Cardiac surgery | 10 years (at the end of study)
  Percentage of patients requiring cardiac surgery for the cardiac carcinoid heart disease
5HIAA levels | 10 years (at the end of study)
  Correlation between urinary 5HIAA levels at diagnosis and occurrence of carcinoid heart disease
Survival | 10 years (at death or at the end of study)
  Overall survival in patents with and without carcinoid heart disease

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CHU Bordeaux - Hopital Haut-Lévèque, Bordeaux
  - APHP Beaujon, Clichy
  - CHU Dijon, Dijon
  - GHICL Lille, Lille
  - Centre Oscar Lambret, Lille
  - CHRU Lille, Lille
  - Hôpital Edouard HERRIOT, Institut du Cancer - Hospices Civils de Lyon, Lyon
  - Institut Paoli-Calmettes, Marseille
  - APHP - Hopital Cochin, Paris
  - APHP - Saint Antoine, Paris
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - Hôpital Haute Pierre, Strasbourg
  - CHU Rangueil, Toulouse
  - CHRU Tours, Tours
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No